CLINICAL TRIAL: NCT00470795
Title: A Randomized, Placebo/Sham-Controlled, Double-Blind Crossover Study to Assess the Efficacy of Acupuncture in the Treatment of Diabetic Gastroparesis.
Brief Title: Acupuncture for Diabetic Gastroparesis
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Protocol to be re-designed (primary outome still GCSI)
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Noah Samuels, Shaare Zedek Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ACP.GP.07
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Diabetic Gastroparesis
Keywords: diabetes; gastroparesis; acupuncture; symptoms; gastric emptying
MeSH Terms: conditions — Diabetes Mellitus; Gastroparesis | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Acupuncture - 2 treatments weekly, 4 weeks (8 treatment)
  Interventions: Other: Acupuncture
- B (Placebo Comparator): Placebo/sham treatment; twice weekly for 4 weeks (total 8 treatments)
  Interventions: Procedure: placebo/sham acupuncture

INTERVENTIONS:
Other: Acupuncture — acupuncture treatment (or placebo), 20 minute treatment each; twice weekly for four weeks (total of eight treatments). repeat treatment schedule following crossover (placebo-treatment)
  Arms: A
Procedure: placebo/sham acupuncture — acupuncture at sham points without skin penetration
  Arms: B

SUMMARY:
Gastroparesis is a common complication of prolonged diabetes mellitus, both with Type 1 and Type 2 forms. Treatment of diabetic gastroparesis ranges from changing dietary habits to medications and invasive procedures, all of which offer only partial and transient relief, with some options having potentially harmful effects. Acupuncture is an ancient treatment which has been found to be beneficial for many ailments, including those involving the gastrointestinal tract. We propose to evaluate whether acupuncture is an effective and safe treatment for diabetic gastroparesis using a randomized, double-blind, placebo/sham-controlled crossover trial. Because symptoms of gastroparesis do not correlate well with objective tests of gastric emptying (i.e., scintigraphy or 13C breath tests), our primary outcome value will be the Gastroparesis Cardinal Symptom Index (GCSI), a reliable and validated instrument for quantifying symptoms in these patients. As a secondary outcome we will measure gastric emptying using a C13-acetate breath test, as well as the SF-12 Short Form Health Survey. Blinding of the participants will be evaluated using a Validation of Blinding Questionnaire at the end of the treatment period.

Diabetic patients suffering from moderate gastroparesis (total GCSI score > 2.50) who fulfill the inclusion criteria (and none of the exclusion criteria) will be eligible to participate in the study. On induction, participants will fill out the GCSI questionnaire and SF-36 survey, and will undergo a C13-acetate breath test. They will then be randomly assigned to either true acupuncture treatment or placebo/sham acupuncture treatment. Each participant will undergo 8 treatments twice-weekly, for a period of 4 weeks. At the end of the eighth treatment session, each participant will again fill out a GCSI questionnaire and SF-12 form, as well as repeating the C13-acetate breath. Following a 4-week washout period, patients will be crossed over to either placebo/sham or true acupuncture treatment, again 8 twice-weekly treatments, for a period of 4 weeks. At the end of the second treatment regimen all participants will again fill out a GCSI questionnaire and SF-12 form, and undergo a C13-acetate breath test. At the end of the second treatment regimen participants will again fill out a Validation of Blinding Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older;
* Controlled diabetes (<250 mg/dL);
* Moderate gastroparesis (GCSI > 2.50);
* Ability to comply with study protocol

Exclusion Criteria:

* Past experience with acupuncture;
* History of gastric surgery, intrapyloric botulinum toxin, gastric pacemaker;
* Uncontrolled diabetes or evidence of diabetic ketoacidosis;
* Malabsorptive syndrome, liver or pulmonary disease;
* Pregnancy or fertility treatments;
* Overt psychopathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
GCSI score | 3 months

SECONDARY OUTCOMES:
SF-12 Health Survey Questionnaire; C-13 acetate breath test | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Noah Samuels, M.D., Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel; Joseph Lysy, M.D., Principal Investigator — Hadassah University Hospital
Locations (2):
- Israel (2):
  - The Center for Integrative Complementary Medicine, Shaare Zedek Medical Center, Jerusalem
  - Dept. of Gastroenterology, Hadassah University Hospital, Jerusalem